CLINICAL TRIAL: NCT02424396
Title: Biological Activity and Safety of Low Dose IL2 in Relapsing Remitting Multiple Sclerosis. Multicentric Randomized Study
Brief Title: Biological Activity and Safety of Low Dose IL2 in Relapsing Remitting Multiple Sclerosis
Acronym: MS-IL2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation ARSEP/AFM (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P130102; 2014-000088-82 (Other: EudractCT)
Record Dates: First submitted 2015-04-20; First posted 2015-04-23 (Estimated); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Interleukin 2, IL2; Relapsing Remitting Multiple Sclerosis; Autoimmune diseases; Regulatory T cells, Tregs
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Autoimmune Diseases | interventions — Interleukin-2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 : IL2 (Experimental): Interleukin-2 (ILT-101)
  Interventions: Drug: IL2
- 2 : Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IL2 — Induction period: repeated administration of low-dose IL-2 Maintenance period: treatment with IL-2
  Arms: 1 : IL2
Drug: Placebo
  Arms: 2 : Placebo

SUMMARY:
Interleukin-2 (IL-2) was initially discovered and used as a stimulator of effector T lymphocytes (Teffs), but is now viewed as a very promising immunoregulatory drug having the capacity to stimulate regulatory T cells (Tregs). At low dose, Il-2 tips the Treg/Teff balance towards Tregs. Recently, it has been shown that Tregs of MS patients have reduced proliferative potential. MS-IL2 will assess the safety and biological efficacy of low-dose IL2 as a Treg inducer in a Relapsing-Remitting Multiple Sclerosis (RRMS), with the aim to stimulate Treg and define potential clinical benefits

DETAILED DESCRIPTION:
In MS-IL2, 30 RRMS patients will be treated in a randomized, double-blind, placebo controlled clinical trial. IL-2 will be administered first as an induction course of IL-2 or placebo each day for 5 days, followed by a maintenance course at the same dose or placebo every two weeks over 6 months.

The primary efficacy criteria will be the % change from baseline in Treg at day-5, which is indicative of the biological response to IL-2.

The secondary efficacy criteria will be (i) the maintenance of regulatory T cells during the 6 months of treatment with IL-2 vs. placebo and (ii) the stabilization or regression of the disease as determined by disease activity parameters assessed by MRI (cumulative number of new lesions in T1 enhanced by gadolinium after 6 months) in the groups treated with IL-2 compared to placebo.

Expected impact: MS-IL2 will define which patient respond to IL2 and which doses prevent relapses in RRMS. In addition, the deep phenomics studies will further provide the foundation for a clinical phase II to define clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years old ;
* Male and Female;
* Presenting relapsing remitting multiple sclerosis as determined by revised McDonald criteria (2010) ;
* On MRI : 1) Presenting 1-2 lesions enhanced by gadolinium (Gd+) (T1) without clinical expression of the disease clinique upon inclusion or 6 months prior to inclusion or 2) presenting one new lesion T2
* Expanded Disability Status Scale (EDSS) score comprised between 0 and 6;
* No flare (with or without any corticosteroid therapy) for the past 2 months
* Under β-Interferon treatment for ≥ 6 months ; or any other first-line treatment of the Relapsing-Remitting Multiple Sclerosis (RRMS): Dimethyl fumarate or teriflunomide treatment for ≥ 6 months or glatiramer acetate for ≥ 9 months
* For women of childbearing age, contraception for more than 2 weeks upon confirmation of inclusion criteria and negative Beta HCG on inclusion visit (D-30 to D-7);
* Patient informed consent should be signed by the patient and investigator before performing any clinical examination required for the study.
* Affiliation to the French Social Security Regimen

Exclusion Criteria:

* Number of lesions enhanced by gadolinium (Gd+) on MRI in T1 > 2 upon inclusion;
* Known intolerance to IL2 (see SPC):

  * Hypersensibility to active substance or one of the excipients ;
  * Signs of evolving infection requiring treatment
  * Other clinically significant chronic disorders (beside RR-MS)
  * History of organ allograft
* Administration of a non-authorized treatment; bolus of corticosteroids in the last 2 months, or treatment with cyclophosphamide, mitoxantrone, or rituximab in the last 6 months;
* Heart failure (≥ grade III NYHA), renal insufficiency, or hepatic insufficiency (transaminase>5N), or lung failure
* White blood cell count <3000 /mm3, lymphocytes< 1000 /mm3, platelets <150 000 /mm3
* Poor venous access not allowing repeated blood tests
* Vaccination with live attenuated virus in the months preceding the inclusion or planned during the study
* Surgery with general anaesthesia during the last 2 months or surgery planned during the study
* Participation in other biomedical research in the last one month or planned during the study
* Concomitant psychiatric disease or any other chronic illness or drug-abuse that could interfere with the ability to comply with the protocol or to give informed consent
* Cancer or history of cancer cured for less than five years (except in situ carcinoma of the cervix or basocellular carcinoma)
* Pregnant or lactating women;
* Men and women of childbearing potential without effective contraception for the duration of treatment
* Patients under a measure of legal protection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-06-13 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2020-06-15 (Actual)

PRIMARY OUTCOMES:
Treg response to low dose IL2 induction course period, expressed as % of total CD4 cells | at day5

SECONDARY OUTCOMES:
Change in Treg percentage on D15 after induction (D1-D5) compared to baseline | at day15
Change in Treg percentage from D15 to M6 compared to baseline | Day 15 to Day 169
The cumulative number of new lesions enhanced by Gd+ (Sum of Gd + lesions on T1 MRI on M2, M4 and M6) | Day 57, Day 113 and Day 169
Frequency of patients free of Gd+ lesions at M6 | Day 169
The cumulative number of new T2 lesions | Day 169
Annual relapse rate (number of relapses observed over a 6 month period) | Day 169
% of patients with flare | Day 169
% of disease free patient i.e % of patient with no clinical symptoms and no activity on MRI | Day 169

CONTACTS AND LOCATIONS:
Overall Officials: David Klatzmann, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (3):
- France (3):
  - Centre d'investigation Clinique - Pitié salpêtrière, Paris
  - Centre d'investigation clinique Biothérapie Immunologie (CIC-BTi) - Groupe Hospitalier Pitié-Salpêtrière - AP-HP, Paris
  - Département des maladies du système nerveux et Centre d'investigation clinique - Groupe Hospitalier Pitié-Salpêtrière - AP-HP, Paris

REFERENCES:
- [Derived] Louapre C, Rosenzwajg M, Golse M, Roux A, Pitoiset F, Adda L, Tchitchek N, Papeix C, Maillart E, Ungureanu A, Charbonnier-Beaupel F, Galanaud D, Corvol JC, Vicaut E, Lubetzki C, Klatzmann D. A randomized double-blind placebo-controlled trial of low-dose interleukin-2 in relapsing-remitting multiple sclerosis. J Neurol. 2023 Sep;270(9):4403-4414. doi: 10.1007/s00415-023-11690-6. Epub 2023 May 28. PMID 37245191